CLINICAL TRIAL: NCT05287217
Title: Post-operative Pain Control With Acetaminophen and Ibuprofen After Functional Endoscopic Sinus Surgery for Chronic Rhinosinusitis: a Prospective Study.
Brief Title: Post-operative Pain Control With Acetaminophen and Ibuprofen After Functional Endoscopic Sinus Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not proceeding this study. Research is not longer relevant
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-1249
Record Dates: First submitted 2022-02-01; First posted 2022-03-18 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Chronic Rhinosinusitis (Diagnosis)
Keywords: Pain Control
MeSH Terms: conditions — Disease; Agnosia | interventions — Analgesia

STUDY DESIGN:
Intervention Model Description: Adult patients will be screened and consented. Group assignment will be determined on an alternating basis. After FESS surgery patients will be given post-operative pain management instructions according to group assignment. Group 1 will take 650mg of acetaminophen every 6 hours and 600mg of ibuprofen every 8 hours for 10 consecutive days after surgery regardless of whether they experience pain or not. Group 2 will take the 650mg of acetaminophen every 6 hours and 600mg of ibuprofen every 8 hours for 10 days after surgery only when needed to control pain. Patients in both groups will record post-operative pain medications for 10 consecutive days after surgery and their level of pain once per day. The patients' post-op follow-up visit will occur 10-14 days after surgery. Medications prescribed for this study are standard of care following FESS surgery. The instructed use of the medications following surgery are being done strictly for comparative and research purposes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Scheduled pain control (Active Comparator): Group 1 patients will be instructed to take 650mg of acetaminophen every 6 hours and 600mg of ibuprofen every 8 hours for 10 consecutive days after surgery regardless of whether they experience pain or not.
  Interventions: Other: Comparison of medication administration for pain control
- Group 2: Pain control as needed. (Active Comparator): Group 2 patients will be instructed to take the 650mg of acetaminophen every 6 hours and 600mg of ibuprofen every 8 hours for 10 days after surgery only when needed to control pain.
  Interventions: Other: Comparison of medication administration for pain control

INTERVENTIONS:
Other: Comparison of medication administration for pain control — Measuring pain control following FESS surgery

SUMMARY:
The safest and most effective post-operative pain control regimen after functional endoscopic sinus surgery (FESS) has been the subject of persistent research. This prospective study will compare post-operative pain control when managed either by a defined medication schedule or medication taken on an as-needed basis after functional endoscopic sinus surgery for chronic rhinosinusitis.

Prior to surgery, patients will be randomly selected to be in one of two treatment arms. One group will receive instructions to take specific medications (acetaminophen and ibuprofen on a specific schedule post-operatively. The second treatment groups will be instructed to take the same medications but on an as needed basis for pain. Patients will also be provided with an option of a limited supply of narcotic analgesics for pain should they be needed.

Post-operative pain control will be assessed by the patient with a pain-diary documenting perceived levels of pain for 10 days post-operatively using a validated visual analog scale. At the conclusion of the study the records of medications taken along with pain responses will be compared between groups

DETAILED DESCRIPTION:
The safest and most effective post-operative pain control regimen after functional endoscopic sinus surgery (FESS) has been the subject of persistent debate and research for many years. The main reasons for this debate is due to two factors: 1) endoscopic sinus surgery is a commonly performed as an outpatient procedure by both generalist and sub-specialized Otolaryngologists. Therefore, there is limited controlled data on pain levels and pain control post-surgery. 2) The ongoing opiate crisis in the United States raises concern of over-prescribing narcotic pain medication post-surgery when it is not necessary.

Of the 600,000 ambulatory sinonasal procedures performed annually in the United States, over 255,000 are sinus surgeries.1 Coupled with an estimated 2 million Americans suffering from opioid use disorders, there is a necessity for further research into minimizing the use of opioids for pain management as well as for testing non-opioid pain management options for postoperative FESS patients.

This study builds on prior research studying optimal non-narcotic analgesia after FESS. A 2018 survey by the American Rhinologic Society showed that over 90% of responders prescribed at least one type of opioid for postoperative pain after FESS. While the majority of Otolaryngologists routinely prescribe opioids, several studies have demonstrated that acetaminophen and NSAIDs can be just as effective in managing postoperative pain in FESS patients. Despite prior concerns that ibuprofen increases risk of epistaxis after FESS, it has been shown that bleeding complications following FESS are negligible.

Recent literature in other surgical sub-specialties has shown that scheduled non-narcotic pain medication significantly reduced patient's post-operative pain scores as compared to those taking it on an as-needed basis.6 In Otolaryngology, the practice of scheduled acetaminophen and ibuprofen has been documented to reduce admissions due to post-tonsillectomy pain.7 Despite the rising trend of non-narcotic pain regimens after surgery, the most appropriate method for instituting this in FESS patients has only been briefly evaluated. A 2006 study showed that scheduled medication use versus as-needed modified-release acetaminophen allowed patients to return to normal daily activities more rapidly and with less pain than patients taking post-operative pain medications on an as needed basis. However, this pain regimen did not include NSAIDs, and modified release acetaminophen is not commonly available in the United States.

This study will evaluate post-operative pain management in patients undergoing outpatient functional endoscopic sinus surgery. Patients will be randomized into one of two study groups: Group 1: Patients instructed to follow a predetermined post-operative acetaminophen and ibuprofen medication schedule, and Group 2: patients instructed to take acetaminophen and ibuprofen as needed after the onset of pain/discomfort. Additionally, all patients in both study groups will be provided a limited number of narcotic pills (Norco) for pain. Patients will be advised to only take the pills for pain that is not controlled by the post-operative acetaminophen and ibuprofen medications.

Pain control will be self-assessed by each patient for the first 10 days after surgery using a validated visual-analog scale (VAS).

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥18 years of age.
* Patients of the PI (Dr. Joe) scheduled for sinus surgery at UI Health.
* Patients with CRS defined as greater than 12 weeks of 2 of the 4 following symptoms: nasal obstruction/congestion, mucopurulent discharge (nasal or postnasal), facial pain/pressure, or decreased/loss of smell + endoscopic/radiographic evidence of disease.
* CRS patients with or without nasal polyps.
* Patients who are COVID-19 negative.
* Patients that understand the purpose and procedures of the study and who agree to participate.
* Patients who have the capacity to consent autonomously.

Exclusion Criteria:

* Males and females < 18 years of age.
* Patients of the PI (Dr. Joe) who are not scheduled for sinus surgery at UI Health.
* Patients who do not have CRS.
* Patients who have allergies to acetaminophen, ibuprofen, and related non-steroidal anti-inflammatory drugs (NSAIDS).
* Patients with kidney or liver dysfunction, cirrhosis, metabolic deficiencies, inflammatory bowel disease, peptic ulcer disease, chronic malnutrition, who have had a previous skull base surgery, or who are currently undergoing cancer treatment.
* Woman who are pregnant or breastfeeding will be excluded.
* Patients with a history of drug and/or narcotic abuse will be excluded.
* COVID-19 positive patients.
* Patients who are not able to understand the purpose and procedures of the study and who do not wish to participate.
* Patients that do not have the capacity to consent autonomously.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-07-29 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Scheduled versus as needed pain management following FESS surgery | 10 days
  The primary outcome measure will compare patient self-assessed pain levels, between the 2 study groups, using a Faces Pain Scale Record. The faces pain scale ranges from 0 to 10 with 0 being no pain and 10 being worst possible pain. Each number on the scale is associated with a pain description and an animated face associated with the description.

SECONDARY OUTCOMES:
Does scheduled pain management decrease narcotic use. | 10 days
  The second outcome measure will quantify (count) the number of narcotic (Norco) pills taken by each patient post-operatively in the 2 study groups.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Joe, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Department of Otolaryngology-Head and Neck Surgery, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bhattacharyya N. Ambulatory sinus and nasal surgery in the United States: demographics and perioperative outcomes. Laryngoscope. 2010 Mar;120(3):635-8. doi: 10.1002/lary.20777. PMID 20058315
- [Background] [2] Substance Abuse and Mental Health Services Administration. (2019). Key substance use and mental health indicators in the United States: Results from the 2018 National Survey on Drug Use and Health (HHS Publication No. PEP19-5068, NSDUH Series H-54). Rockville, MD: Center for Behavioral Health Statistics and Quality, Substance Abuse and Mental Health Services Administration. Retrieved from https://www.samhsa.gov/data/
- [Background] Gray ML, Fan CJ, Kappauf C, Kidwai S, Colley P, Iloreta AM, Govindaraj S. Postoperative pain management after sinus surgery: a survey of the American Rhinologic Society. Int Forum Allergy Rhinol. 2018 Oct;8(10):1199-1203. doi: 10.1002/alr.22181. Epub 2018 Jul 18. PMID 30019397
- [Background] Nguyen KK, Liu YF, Chang C, Park JJ, Kim CH, Hondorp B, Vuong C, Xu H, Crawley BK, Simental AA, Church CA, Inman JC. A Randomized Single-Blinded Trial of Ibuprofen- versus Opioid-Based Primary Analgesic Therapy in Outpatient Otolaryngology Surgery. Otolaryngol Head Neck Surg. 2019 May;160(5):839-846. doi: 10.1177/0194599819832528. Epub 2019 Mar 5. PMID 30832548
- [Background] Wu AW, Walgama ES, Genc E, Ting JY, Illing EA, Shipchandler TZ, Higgins TS. Multicenter study on the effect of nonsteroidal anti-inflammatory drugs on postoperative pain after endoscopic sinus and nasal surgery. Int Forum Allergy Rhinol. 2020 Apr;10(4):489-495. doi: 10.1002/alr.22506. Epub 2019 Dec 13. PMID 31834679
- [Background] Poljak D, Chappelle J. The effect of a scheduled regimen of acetaminophen and ibuprofen on opioid use following cesarean delivery. J Perinat Med. 2020 Feb 25;48(2):153-156. doi: 10.1515/jpm-2019-0322. PMID 31951589
- [Background] Shelton FR, Ishii H, Mella S, Chew D, Winterbottom J, Walijee H, Brown R, Chisholm EJ. Implementing a standardised discharge analgesia guideline to reduce paediatric post tonsillectomy pain. Int J Pediatr Otorhinolaryngol. 2018 Aug;111:54-58. doi: 10.1016/j.ijporl.2018.05.020. Epub 2018 May 19. PMID 29958614
- [Background] Kemppainen TP, Tuomilehto H, Kokki H, Seppa J, Nuutinen J. Pain treatment and recovery after endoscopic sinus surgery. Laryngoscope. 2007 Aug;117(8):1434-8. doi: 10.1097/MLG.0b013e3180600a16. PMID 17572643
- [Background] Gao Y, Wang C, Wang G, Cui X, Yang G, Lou H, Zhang L. Benefits of Enhanced Recovery After Surgery in Patients Undergoing Endoscopic Sinus Surgery. Am J Rhinol Allergy. 2020 Mar;34(2):280-289. doi: 10.1177/1945892419892834. Epub 2019 Dec 4. No abstract available. PMID 31799861
- [Background] Svider PF, Nguyen B, Yuhan B, Zuliani G, Eloy JA, Folbe AJ. Perioperative analgesia for patients undergoing endoscopic sinus surgery: an evidence-based review. Int Forum Allergy Rhinol. 2018 Jul;8(7):837-849. doi: 10.1002/alr.22107. Epub 2018 Apr 12. PMID 29645361
- [Background] Du E, Farzal Z, Stephenson E, Tanner A, Adams K, Farquhar D, Weissler M, Patel S, Blumberg J, Jowza M, Hackman T, Zanation A. Multimodal Analgesia Protocol after Head and Neck Surgery: Effect on Opioid Use and Pain Control. Otolaryngol Head Neck Surg. 2019 Sep;161(3):424-430. doi: 10.1177/0194599819841885. Epub 2019 Apr 9. PMID 30961428
- [Background] Oltman J, Militsakh O, D'Agostino M, Kauffman B, Lindau R, Coughlin A, Lydiatt W, Lydiatt D, Smith R, Panwar A. Multimodal Analgesia in Outpatient Head and Neck Surgery: A Feasibility and Safety Study. JAMA Otolaryngol Head Neck Surg. 2017 Dec 1;143(12):1207-1212. doi: 10.1001/jamaoto.2017.1773. PMID 29049548
- [Background] Bijur PE, Silver W, Gallagher EJ. Reliability of the visual analog scale for measurement of acute pain. Acad Emerg Med. 2001 Dec;8(12):1153-7. doi: 10.1111/j.1553-2712.2001.tb01132.x. PMID 11733293
- [Background] Ferreira-Valente MA, Pais-Ribeiro JL, Jensen MP. Validity of four pain intensity rating scales. Pain. 2011 Oct;152(10):2399-2404. doi: 10.1016/j.pain.2011.07.005. PMID 21856077